CLINICAL TRIAL: NCT00637624
Title: A Randomized Double-blind Study of N-AcetylCysteine vs. Placebo to Prevent Neurotoxicity Induced by Platinum Containing Chemotherapy in Patients Treated for (Non)Small Cell Lung Cancer and Malignant Mesothelioma
Brief Title: N-AcetylCysteine vs. Placebo to Prevent Neurotoxicity Induced by Platinum Containing Chemotherapy
Acronym: NAC-PNP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit enough patients
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LTC-510-100108-Bahce; CCMO: NL19614.091.07; EudraCT: 2007-002787-95
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Small Cell Lung; Mesothelioma
Keywords: Acetylcysteine; Cisplatin; Neuropathy; Antioxidants
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Mesothelioma | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): N-Acetylcysteine
  Interventions: Drug: N-Acetylcysteine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-Acetylcysteine — N-Acetylcysteine intravenously once every 3 weeks 40 mg/kg
  Other Names: Fluimucil
  Arms: 1
Drug: Placebo — Placebo once every 3 weeks intravenous saline fluid
  Arms: 2

SUMMARY:
In this study we want to investigate the efficacy of N-acetylcysteine (NAC), which is an anti-oxidant, in the prevention of cisplatin-induced neural toxicity, in patients treated for lung cancer with chemotherapy containing cisplatin.

DETAILED DESCRIPTION:
Background of the study:

Cisplatin (CDDP) is a major compound in chemotherapy in patients with non-small cell lung cancer (NSCLC), small cell lung cancer (SCLC) and malignant mesothelioma. Cisplatin is associated with a number of side-effects, one of which is neurotoxicity. For a number of patients this neurotoxicity is a dose-limiting side-effect. At this point no measures are taken to prevent the occurrence of neurotoxicity during treatment with cisplatin. Recent studies have shown that the association of anti-oxidants to the treatment with cisplatin has a neuroprotective effect without loss of anti-tumour efficacy of cisplatin. One of these anti-oxidants is glutathione (GSH), this is a natural anti-oxidant that is synthesized in all cells, mainly in the liver and the muscles. This GSH plays a central role in the pathophysiology (of efficacy and of side-effects) of cisplatin. We want to investigate the efficacy of N-acetylcysteine (NAC), which serves as a substrate for the synthesis of GSH, in the prevention of cisplatin-induced neurotoxicity.

Objective of the study:

* The primary objective is to establish the neuroprotective efficacy of NAC against cisplatin-induced neurotoxicity. Mainly the sensory neuronal guidance will be assessed before and after treatment with cisplatin in a group of patients receiving NAC compared to a control-group receiving placebo. If peripheral neuropathy can't be measured, neuropathy will be assessed as ototoxicity through measuring audiograms.
* The secondary objectives are establishing the protective effect of NAC regarding other cisplatin-induced side-effects such as haematological pathology (anaemia, leucopenia, thrombopenia, febrile neutropenia), loss of creatinine clearance and occurrence of liver-chemistry abnormalities. Secondary objectives include also establishing the effect on tumour response, clinical performance (Karnofsky performance index) and quality of life.

Study design:

Monocenter, non-academical teaching hospital, double-blind randomized placebo-controlled study.

Study population:

50 Consecutive patients, who will receive at least 4 cycles of cisplatin in the treatment of NSCLC, SCLC and malignant mesothelioma, will be admitted, irrespective of the disease stage.

Intervention:

Patients will be randomized in a placebo-arm and a NAC-arm. They will receive study-medication (NAC or placebo) intravenously every 3 weeks, each time 6 hours after the completion of the cisplatin-infusion.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

* Burdens: Patients will have to undergo three electromyographic (EMG) tests, which will normally take place during the course of the whole treatment, therefore patients will have to visit the hospital to be measured. To minimize this burden, the EMG-measurements will be planned on the same day, the patient has to visit the hospital for reasons regarding his/her regular chemotherapy-treatment. Only surface patch electrodes will be used (no needle electrodes). All other information will be obtained from the patients' files (blood samples, physic evaluations, etc) these are considered to be part of the routines of treatment. When EMG's can not be measured, audiograms will be used, these audiograms are also part of the routines of treatment, so are not considered an extra burden. Patients will have to fill in Quality of Life questionnaires.
* Risks: NAC is a well known drug, used for over thirty years, that is well tolerated. For intravenous NAC, allergic reactions have been reported. There is also a theoretical risk, that NAC may reduce anti-tumour efficacy of cisplatin, this risk will be theoretically ruled out by appropriate dosing of NAC. After inclusion of the first 30 patients an interim analysis will be performed regarding the tumour response.
* Benefits: NAC will possibly prevent the occurrence of neurotoxicity, improving quality of life. This may, in turn, result in less probability of dose-reductions and of preterm arrest of treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnose is histologically or cytologically proven (NSCLC,SCLC), malignant mesothelioma (histologically)
* at least 4 cycles of cisplatin are planned
* adequate renal function (creatinine clearance as calculated by Cockroft-Gault method > 60 ml/min)
* Karnofsky performance score > 60 %
* written informed consent
* patient must be able to comply with study measurements i.e. hospital visits for EMG and QoL assessments
* age ≥ 18 years

Exclusion Criteria:

* patients with pre-existing neuropathy
* patients not willing to stop earlier prescribed NAC
* patients not willing to stop vitamins E and A above daily advisory dosage
* uncontrolled metastasis in the central or peripheral nervous system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
The occurrence of peripheral neuropathy: with the peripheral neuropathy score (PNP-score) and the electrophysiological measurements. If no EMG is available, then audiometric measurements will be taken into account. | 5 months

SECONDARY OUTCOMES:
haematological abnormalities | 5 months
creatinine clearance. | 5 months
liver chemistry abnormalities | 5 months
Karnofski Performance Score | 5 months
Quality of life | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Idris Bahce, MD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands